CLINICAL TRIAL: NCT04432896
Title: Systemic Nickel Allergy Syndrome: Intervention Study for the Assessment of the Dietary Indications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Hellas Cena, Prof, University of Pavia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17042020
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Nickel Sensitivity; Allergy; Nickel; Eczema; Women; Systemic Syndrome
Keywords: women; Systemic syndrome; Nickel Allergy
MeSH Terms: conditions — Hypersensitivity; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New dietary protocol (Experimental): Exclusion of food containing nickel (duration: 4 weeks) + gradual weekly reintroduction of food containing nickel (duration: 4 weeks) under the supervision of a trained dietician who monitors symptoms related to systemic nickel allergy syndrome.
  Interventions: Other: Dietary protocol
- Traditional dietary protocol (Active Comparator): Exclusion of foods containing nickel without monitoring for symptoms related to systemic nickel allergy syndrome by a trained dietician.
  Interventions: Other: Dietary protocol

INTERVENTIONS:
Other: Dietary protocol — Dietary protocol to manage symptoms related to Systemic Nickel Allergy Syndrome.

SUMMARY:
Background: Nickel is a silvery metal widely used in nature and contained in many foods. Exposure to nickel is responsible for two different types of adverse reactions: Allergic Contact Dermatitis (DAC) and Systemic Nickel Allergy Syndrome (SNAS). The latter is characterized by the presence of extra-cutaneous manifestations, in addition to the skin lesions of the DAC, related to the introduction of nickel-containing foods. Therefore, a nutritional intervention is essential to reduce the symptoms of SNAS. Currently in the literature there are no nutritional guidelines on the treatment and management of patients suffering from SNAS and often the indications provided to patients involve the exclusion of groups of foods for prolonged periods, with the consequent risk of developing nutritional deficiencies and malnutrition.

Objectives: to evaluate the efficacy of dietary indications, developed on the most recent scientific evidence, useful for the management of the symptoms associated with adverse reactions to Nickel. Provide practical indications to specialist staff in multidisciplinary patient management and make the patient aware of his problem and help him understand how to manage it independently.

Target population: subjects over the age of 18, female, belonging to the U.O. Occupational Medicine Allergology Section at ICS Maugeri of Pavia, with previous diagnosis of Nickel allergy (patch test) and with the presence of gastrointestinal symptoms related to allergy.

DETAILED DESCRIPTION:
The primary objective of this intervention study is the evaluation of the efficacy of dietary indications, developed on the most recent scientific evidence, useful for the management of the symptoms associated with adverse reactions to nickel.

The secondary objective is to:

* verify the correlation between the consumption of a specific food and the onset of gastroenteric symptoms;
* provide a practical indication to the dietician who acts in concert with the figure of the dietician and allergist in the multidisciplinary management of the patient in order to manage and contain the symptoms;
* make the patient aware of his problem and help him understand how to manage it autonomously, from a food point of view, thus promoting a diet as complete and balanced as possible and at the same time reduce the risk of nutritional deficiencies, such as deficits of minerals and vitamins, and the consequent impact on the state of health.

In this experimental study, each patient will be assessed at the baseline time (T0) in which the pathological and physiological history and anthropometric data (weight, height, waist circumference, BMI) will be collected.The patients of the intervention group will be given dietetic indications by the reference dietitian, which must be followed for 8 weeks. In short, the indications provide for an exclusion period (4 weeks). At the end of this phase (T1) one group of foods per week will be reintroduced on the basis of their nickel content.The reintroduction will begin with the group of foods with a lower nickel content and will proceed gradually for a period of 4 weeks (T1a, T1b, T1c, T2). In order to monitor the trend of gastroenteric symptoms, a diary of symptoms will be administered at baseline time (T0) which must be completed for the duration of the study (T1a, T1b, T1c, T2) and which will be delivered and evaluated by the dietician and the reference clinician. To ensure adequate patient support and to monitor compliance with the indications provided, the referring dietitian will have to contact individual patients once a week by telephone or e-mail.

ELIGIBILITY:
Inclusion Criteria:

* patients on first access aged 18 or over;
* nickel phosphate sensitized patients (patch test: ++ or +++);
* monosensitized or polisensitized patients;
* patients with the presence of allergic gastrointestinal symptoms;
* patients negative to diagnostic tests for other allergies;
* signature of informed consent.

Exclusion Criteria:

* patients positive for diagnostic tests for other allergies;
* polysensitized patients with additives and preservatives, to exclude any confounding effects;
* patients who have previously received dietary indications for allergy management;
* patients who have been diagnosed with IBD (Irritable Bowel Disease) such as Ulcerative Rectocolitis, Chron's disease, IBS;
* patients in whom a Eating and Nutrition Disorder (DAN) has been diagnosed;
* patients with malignancies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
protocol nickel free | 2 years
  to evaluate the efficacy of dietary indications, developed on the most recent scientific evidence, useful for the management of the symptoms associated with adverse reactions to nickel.
  Throughout the study: therefore during the first phase in which a nickel free diet is followed and during the second phase of gradual reintegration of food containing nickel, patients must fill in a diary of what they eat weekly. The efficacy of dietary indications is evaluated using the visual analog scale. Both the symptoms related to the gastro intestinal system (nausea, diarrhea, vomiting, bloating of the intestine), and those extra intestinal such as headache, itching are evaluated.

SECONDARY OUTCOMES:
Nickel free diet and symptoms | 2 years
  verify the correlation between the consumption of a specific food and the onset of gastroenteric symptoms, using a dietary in wich the patien described what they eat and their specific symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No